CLINICAL TRIAL: NCT03643276
Title: International Collaborative Treatment Protocol for Children and Adolescents With Acute Lymphoblastic Leukemia - AIEOP-BFM ALL 2017
Brief Title: Treatment Protocol for Children and Adolescents With Acute Lymphoblastic Leukemia - AIEOP-BFM ALL 2017
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Martin Schrappe (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Sponsor-Investigator, Martin Schrappe, Professor MD, FRCP (Glasg), Chair of Pediatrics I, University Hospital Schleswig-Holstein
Organization: University Hospital Schleswig-Holstein (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: AIEOP-BFM ALL 2017
Record Dates: First submitted 2018-07-12; First posted 2018-08-22 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric
Keywords: Acute Lymphoblastic Leukemia; Childhood; Pediatric; Immunotherapy; Blinatumomab; Proteasome Inhibitor; Bispecific antibody; Bortezomib; Chemotherapy; Randomized trial
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab; Bortezomib; Cyclophosphamide; Cytarabine; Daunorubicin; Doxorubicin; Dexamethasone; Etoposide; fludarabine phosphate; Ifosfamide; Mercaptopurine; Methotrexate; pegaspargase; Prednisolone; Prednisone; Thioguanine; Vincristine; Vindesine; Asparaginase

STUDY DESIGN:
Intervention Model Description: pB-ALL/MR: 2 parallel groups (R-MR) or 2x2 factorial design (R-eHR, R-MR) depending on early risk group assignment.
  pB-ALL/HR: 2 parallel groups (R-HR) or 2x2 factorial design (R-eHR, R-HR) depending on early risk group assignment.
  T-ALL/early non-SR: 2 parallel groups (R-T).
  pB-ALL/SR: Single group.
  T-ALL/early SR: Single group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- pB: early (non-)HR-standard/MR-standard (Active Comparator): Induction (5 wks): "Protocol IA" with prednisolone, vincristine, daunorubicin, pegaspargase, IT methotrexate (MTX)
  Consolidation (6 w/4 w): "Consolidation extended" (control arm of randomization R-eHR) with cyclophosphamide, cytarabine, 6-mercaptopurine (6-MP), IT MTX, dexamethasone, vincristine, pegaspargase or "Consolidation short" (standard arm of early non-HR group) with cyclophosphamide, cytarabine, 6-mercaptopurine, IT MTX
  Extra-compartment phase (8 wks): "Protocol M" with 6-MP, HD-MTX, IT MTX
  Reinduction (6 wks): "Protocol II" with dexamethasone, vincristine, doxorubicin, pegaspargase, IT MTX, cyclophosphamide, tioguanine, cytarabine
  Maintenance (until 2 years after initial diagnosis): 6-MP, MTX [without preceding blinatumomab (control arm of randomization R-MR)]
  Erwinase is given in case of allergy to pegaspargase.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Drug: Doxorubicin; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisolone; Drug: Tioguanin; Drug: Vincristine; Drug: Erwinase
- pB: early HR-exp./MR-standard (Experimental): Induction (5 w): "Protocol IA" with prednisolone, vincristine, daunorubicin, pegaspargase, IT MTX
  Consolidation (6 w): "Consolidation extended+BZM" (experimental arm of randomization R-eHR) with cyclophosphamide, cytarabine, 6-MP, IT MTX, dexamethasone, vincristine, pegaspargase, bortezomib (given at 1.3 mg/m²/dose on days 50, 53, 56 and 59)
  Extra-compartment phase (8 wks): "Protocol M" with 6-MP, HD-MTX, IT MTX
  Reinduction (6 wks): "Protocol II" with dexamethasone, vincristine, doxorubicin, pegaspargase, IT MTX, cyclophosphamide, tioguanine, cytarabine
  Maintenance (until 2 yrs after initial diagnosis): 6-MP, MTX [without preceding blinatumomab (control arm of randomization R-MR)]
  Erwinase is given in case of allergy to pegaspargase.
  Interventions: Drug: Bortezomib; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Drug: Doxorubicin; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisolone; Drug: Tioguanin; Drug: Vincristine; Drug: Erwinase
- pB: early (non)HR-standard/MR-exp. (Experimental): Induction (5 w): "Protocol IA" with prednisolone, vincristine, daunorubicin, pegaspargase, IT MTX
  Consolidation (6 w/4 w): "Consolidation extended" (control arm in randomization R-eHR) with cyclophosphamide, cytarabine, 6-MP, IT MTX, dexamethasone, vincristine, pegaspargase or "Consolidation short" (standard arm of early non-HR group) with cyclophosphamide, cytarabine, 6-mercaptopurine, IT MTX
  Extra-compartment phase (8 w): "Protocol M" with 6-MP, HD-MTX, IT MTX
  Reinduction (6 w): "Protocol II" with dexamethasone, vincristine, doxorubicin, pegaspargase, IT MTX, cyclophosphamide, tioguanine, cytarabine
  Blinatumomab (4 w): 1 cycle blinatumomab given at 15 µg/m²/day for 28 days (experimental arm of randomization R-MR)
  Maintenance (until 2 yrs after initial diagnosis): 6-MP, MTX
  Erwinase is given in case of allergy to pegaspargase.
  Interventions: Drug: Blinatumomab; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Drug: Doxorubicin; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisolone; Drug: Tioguanin; Drug: Vincristine; Drug: Erwinase
- pB: early HR-exp./MR-exp. (Experimental): Induction (5 w): "Protocol IA" with prednisolone, vincristine, daunorubicin, pegaspargase, IT MTX
  Consolidation (6 w): "Consolidation extended+BZM" (experimental arm of randomization R-eHR) with cyclophosphamide, cytarabine, 6-MP, IT MTX, dexamethasone, vincristine, pegaspargase, bortezomib (given at 1.3 mg/m²/dose on days 50, 53, 56 and 59)
  Extra-compartment phase (8 w): "Protocol M" with 6-MP, HD-MTX,IT MTX
  Reinduction (6 weeks): "Protocol II" with dexamethasone, vincristine, doxorubicin, PEG-L-asparaginase, IT MTX, cyclophosphamide, tioguanine, cytarabine
  Blinatumomab (4 w): 1 cycle blinatumomab given at 15 µg/m²/day for 28 days (experimental arm of randomization R-MR)
  Maintenance phase (until 2 yrs after initial diagnosis): 6-MP, MTX
  Erwinase is given in case of allergy to pegaspargase.
  Interventions: Drug: Blinatumomab; Drug: Bortezomib; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Drug: Doxorubicin; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisolone; Drug: Tioguanin; Drug: Vincristine; Drug: Erwinase
- pB: early (non-)HR-standard/HR-standard (Active Comparator): Induction (5 w): as in other pB arms
  Consolidation (6 w/4 w): "Consolidation extended" (control arm in randomization R-eHR) with cyclophosphamide, cytarabine, 6-MP, IT methotrexate, dexamethasone, vincristine, pegaspargase or "Consolidation short" (standard arm of early non-HR group) with cyclophosphamide, cytarabine, 6-MP, IT MTX
  Intensified consolidation (3x5 d): Block HR-1' followed by HR-2' and HR-3' (control arm in randomization R-HR) with dexamethasone, vincristine, vindesine, daunorubicin, HD-MTX, IT MTX, HD-cytarabine, cyclophosphamide, ifosfamide, pegaspargase, etoposide
  Reinduction (3x4 w): "Protocol III" given 3 times with dexamethasone, vincristine, doxorubicin, pegaspargase, IT MTX, cyclophosphamide, tioguanine, cytarabine
  Maintenance (until 2 yrs after init. diagnosis): 6-MP, MTX
  Erwinase is given in case pegaspargase allergy. Pts with poor response to intensified consolidation receive Myocet-FLA (Myocet, fludarabine, HD-cytarabine, IT-MTX).
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Myocet; Drug: Dexamethasone; Drug: Doxorubicin; Drug: Etoposide; Drug: Fludarabine Phosphate; Drug: Ifosfamide; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisolone; Drug: Tioguanin; Drug: Vincristine; Drug: Vindesine; Drug: Erwinase
- pB: early HR-exp./HR-standard (Experimental): Induction (5 w): as in other pB arms
  Consolidation (6 w): "Consolidation extended+BZM" (experimental arm of randomization R-eHR) with cyclophosphamide, cytarabine, 6-MP, IT MTX, dexamethasone, vincristine, pegaspargase, bortezomib (1.3 mg/m²/dose on days 50, 53, 56 and 59)
  Intensified consolidation (3x5 d): Block HR-1' followed by HR-2' and HR-3' (control arm in randomization R-HR) with dexamethasone, vincristine, vindesine, daunorubicin, HD-MTX, IT MTX, HD-cytarabine, cyclophosphamide, ifosfamide, pegaspargase, etoposide
  Reinduction (3x4 w): as in arm "pB: early (non-)HR-standard/HR-standard"
  Maintenance (until 2 yrs after initial diagnosis): 6-MP, MTX
  Erwinase is given in case of allergy to pegaspargase. Pts with poor response to intensified consolidation receive Myocet-FLA (Myocet, fludarabine, HD-cytarabine, IT-MTX)
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Myocet; Drug: Dexamethasone; Drug: Doxorubicin; Drug: Etoposide; Drug: Fludarabine Phosphate; Drug: Ifosfamide; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisolone; Drug: Tioguanin; Drug: Vincristine; Drug: Vindesine; Drug: Erwinase
- pB: early (non-)HR-standard/HR-exp. (Experimental): Induction (5 w): as in other pB arms
  Consolidation (6 w/4 w): "Consolidation extended" (control arm in randomization R-eHR) with cyclophosphamide, cytarabine, 6-MP, IT MTX, dexamethasone, vincristine, pegaspargase or "Consolidation short" (standard arm of early non-HR group) with cyclophosphamide, cytarabine, 6-MP, IT MTX
  Intensified consolidation (1x5 d + 2x28 d): Block HR-1' with dexamethasone, vincristine, HD-MTX, IT MTX, HD-cytarabine, cyclophosphamide, pegaspargase followed by 2 cycles blinatumomab at 15 µg/m²/day for 28 days per cycle plus 2x2 doses IT MTX (experimental arm of randomization R-HR)
  Reinduction (3x4 weeks): as in arm "pB: early (non-)HR-standard/HR-standard"
  Maintenance (until 2 yrs after init. diagnosis): 6-MP, MTX
  Erwinase is given in case of pegaspargase allergy. Pts with poor response to intensified consolidation receive Myocet-FLA (Myocet, fludarabine, HD-cytarabine, IT-MTX)
  Interventions: Drug: Blinatumomab; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Myocet; Drug: Dexamethasone; Drug: Doxorubicin; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisolone; Drug: Tioguanin; Drug: Vincristine; Drug: Erwinase
- pB: early HR-exp./HR-exp. (Experimental): Induction (5 w): as in other pB arms
  Consolidation (6 w): "Consolidation extended+BZM" (experimental arm of randomization R-eHR) with cyclophosphamide, cytarabine, 6-MP, IT MTX, dexamethasone, vincristine, pegaspargase, bortezomib (1.3 mg/m²/dose on days 50, 53, 56 and 59)
  Intensified consolidation (1x5 d + 2x28 d): Block HR-1' with dexamethasone, vincristine, HD-MTX, IT MTX, HD-cytarabine, cyclophosphamide, pegaspargase followed by 2 cycles blinatumomab at 15 µg/m²/day for 28 days per cycle plus 2x2 doses IT MTX (experimental arm of randomization R-HR)
  Reinduction (3x4 weeks): as in arm "pB: early (non-)HR-standard/HR-standard" Maintenance (until 2 yrs after initial diagnosis): 6-MP, MTX
  Erwinase is given in case of allergy to pegaspargase. Pts with poor response to intensified consolidation receive Myocet-FLA (Myocet, fludarabine, HD-cytarabine, IT-MTX)
  Interventions: Drug: Blinatumomab; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Myocet; Drug: Dexamethasone; Drug: Doxorubicin; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisolone; Drug: Tioguanin; Drug: Vincristine; Drug: Erwinase
- pB: early non-HR/SR (Other): Induction (5 w): "Protocol IA" with prednisolone, vincristine, daunorubicin, pegaspargase, IT MTX
  Consolidation (4 w): "Consolidation short" with cyclophosphamide, cytarabine, 6-mercaptopurine, IT MTX
  Extra-compartment phase (8 w): "Protocol M" with 6-MP, HD-MTX, IT MTX
  Reinduction (6 w): "Protocol II" with dexamethasone, vincristine, doxorubicin, pegaspargase, IT MTX, cyclophosphamide, tioguanine, cytarabine
  Maintenance (until 2 yrs after initial diagnosis): 6-MP, MTX
  Erwinase is given in case of allergy to pegaspargase.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Drug: Doxorubicin; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisolone; Drug: Tioguanin; Drug: Vincristine; Drug: Erwinase
- T: early non-SR-standard/(non-)HR (Active Comparator): Induction (5 w): "Protocol IA-Dexa" with prednisolone/dexamethasone, vincristine, daunorubicin, pegaspargase, IT MTX or "Protocol IA-CPM" with prednisolone instead of dexamethasone and additional CPM
  Consolidation (4 w): "Protocol IB regular" (control arm in randomization. R-T) with cyclophosphamide, cytarabine, 6-mercaptopurine, IT MTX
  non-HR extra-compartment phase and reinduction: as in arm "pB: early non-HR/SR"
  HR intensified consolidation and reinduction: as in arm "pB: early (non-)HR-standard/HR-standard"
  Maintenance (until 2 yrs after initial diagnosis): 6-MP, MTX
  Erwinase is given in case of allergy to pegaspargase. Pts with poor response to intensified consolidation receive Myocet-FLA (Myocet, fludarabine, HD-cytarabine, IT-MTX)
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Myocet; Drug: Dexamethasone; Drug: Doxorubicin; Drug: Etoposide; Drug: Fludarabine Phosphate; Drug: Ifosfamide; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisolone; Drug: Tioguanin; Drug: Vincristine; Drug: Vindesine; Drug: Erwinase
- T: early non-SR-exp/(non-)HR (Experimental): Induction (5 w): "Protocol IA-Dexa" with prednisolone/dexamethasone, vincristine, daunorubicin, pegaspargase, IT MTX or "Protocol IA-CPM" with prednisolone instead of dexamethasone and additional CPM
  Consolidation (6 w): "Protocol IB long" (experimental arm in randomization R-T) with cyclophosphamide, cytarabine, 6-mercaptopurine, IT MTX
  non-HR extra-compartment phase and reinduction: as in arm "pB: early non-HR/SR"
  HR intensified consolidation and reinduction: as in arm "pB: early (non-)HR-standard/HR-standard"
  Maintenance (until 2 yrs after initial diagnosis): 6-MP, MTX
  Erwinase is given in case of allergy to pegaspargase. Pts with poor response to intensified consolidation receive Myocet-FLA (Myocet, fludarabine, HD-cytarabine, IT-MTX)
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Myocet; Drug: Dexamethasone; Drug: Doxorubicin; Drug: Etoposide; Drug: Fludarabine Phosphate; Drug: Ifosfamide; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisolone; Drug: Tioguanin; Drug: Vincristine; Drug: Vindesine; Drug: Erwinase
- T: early SR/non-HR (Other): Induction (5 w): "Protocol IA-Dexa" with prednisolone/dexamethasone, vincristine, daunorubicin, pegaspargase, IT MTX
  Consolidation (4 w): "Protocol IB regular" with cyclophosphamide, cytarabine, 6-mercaptopurine, IT MTX
  Extra-compartment phase (8 w): "Protocol M" with 6-MP, HD-MTX, IT MTX
  Reinduction (6 w): "Protocol II" with dexamethasone, vincristine, doxorubicin, pegaspargase, IT MTX, cyclophosphamide, tioguanine, cytarabine
  Maintenance (until 2 yrs after initial diagnosis): 6-MP, MTX
  Erwinase is given in case of allergy to pegaspargase.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Drug: Doxorubicin; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisolone; Drug: Tioguanin; Drug: Vincristine; Drug: Erwinase

INTERVENTIONS:
Drug: Blinatumomab — Experimental therapy in randomizations R-HR and R-MR
  Arms: pB: early (non)HR-standard/MR-exp.; pB: early (non-)HR-standard/HR-exp.; pB: early HR-exp./HR-exp.; pB: early HR-exp./MR-exp.
Drug: Bortezomib — Experimental therapy in randomization R-eHR
  Arms: pB: early HR-exp./MR-exp.; pB: early HR-exp./MR-standard
Drug: Cyclophosphamide — Part of standard chemotherapy and included in experimental treatment phase Protocol IB long in randomization R-T
Drug: Cytarabine — Part of standard chemotherapy and included in experimental treatment phase Protocol IB long in randomization R-T and in the intensification block Myocet-FLA for patients with very high relapse risk
Drug: Daunorubicin — Part of standard chemotherapy
Drug: Myocet — Part of intensification block Myocet-FLA for patients with very high relapse risk
  Arms: T: early non-SR-exp/(non-)HR; T: early non-SR-standard/(non-)HR; pB: early (non-)HR-standard/HR-exp.; pB: early (non-)HR-standard/HR-standard; pB: early HR-exp./HR-exp.; pB: early HR-exp./HR-standard
Drug: Dexamethasone — Part of standard chemotherapy
Drug: Doxorubicin — Part of standard chemotherapy
Drug: Etoposide — Part of standard chemotherapy
  Arms: T: early non-SR-exp/(non-)HR; T: early non-SR-standard/(non-)HR; pB: early (non-)HR-standard/HR-standard; pB: early HR-exp./HR-standard
Drug: Fludarabine Phosphate — Part of intensification block Myocet-FLA for patients with very high relapse risk
  Arms: T: early non-SR-exp/(non-)HR; T: early non-SR-standard/(non-)HR; pB: early (non-)HR-standard/HR-standard; pB: early HR-exp./HR-standard
Drug: Ifosfamide — Part of standard chemotherapy
  Arms: T: early non-SR-exp/(non-)HR; T: early non-SR-standard/(non-)HR; pB: early (non-)HR-standard/HR-standard; pB: early HR-exp./HR-standard
Drug: 6-Mercaptopurine — Part of standard chemotherapy and included in experimental treatment phase Protocol IB long in randomization R-T
Drug: Methotrexate — Part of standard chemotherapy
Drug: Pegaspargase — Part of standard chemotherapy
Drug: Prednisolone — Part of standard chemotherapy
  Other Names: Prednisone
Drug: Tioguanin — Part of standard chemotherapy
Drug: Vincristine — Part of standard chemotherapy
Drug: Vindesine — Part of standard chemotherapy
  Arms: T: early non-SR-exp/(non-)HR; T: early non-SR-standard/(non-)HR; pB: early (non-)HR-standard/HR-standard; pB: early HR-exp./HR-standard
Drug: Erwinase — Part of standard chemotherapy as substitute for PEG-L-Asparaginase in case of allergic reaction

SUMMARY:
The understanding of acute lymphoblastic leukemia (ALL) in childhood and adolescence has largely changed due to extensive genetic research in recent years: ALL is now considered to be a very heterogeneous disease group. The leukemia cells present themselves with quite differently activated regulatory mechanisms of the malignant phenotype. The introduction of more accurate methods of assessing therapy response ("minimal residual disease [MRD] tests") has provided new insights into very different mechanisms of action, including factors influenced by host factors; this has had practical clinical consequences for the use of more individualized therapy. Multimodal therapies have enabled a cure level of over 80% for ALL in this age group. However, the own and international study data show that the therapy toxicity of the contemporary chemotherapy concepts has become unacceptably high, in particular with respect to those intensified therapies used for the treatment of patients at high risk of ALL relapse.

The AIEOP-BFM ALL 2017 study therefore aims for an innovative integrated approach that will not only adapt the risk stratification to new prognostic markers using more comprehensive diagnostics, but above all, qualitatively reorient the therapy. The most important consequence will be that this study is testing immunotherapy with the bispecific antibody blinatumomab as an alternative to particularly intensive and toxic chemotherapy elements in precursor B-cell ALL (pB-ALL) patients with detectable chemotherapy resistance and at high risk of relapse. With the aim to complement the effects of the conventional chemotherapy, Blinatumomab is in addition tested in the large group of pB-ALL patients at intermediate relapse risk with seemingly unremarkable leukemia, but who account for a large proportion of all relapses. Targeted therapy is also used in the form of the proteasome inhibitor bortezomib for patients with pB-ALL and slow response to the drugs of the induction chemotherapy with the aim to overcome intrinsic chemotherapy resistance of the ALL cells. In patients with T-lineage ALL, who have particularly poor chances for cure after relapse, the established consolidation chemotherapy has proved to be particularly effective. This chemotherapy phase is therefore tested in a longer and more intensive form in such T-ALL patients with intermediate or slow early treatment response with the aim to reduce the relapses rate in this subgroup.

DETAILED DESCRIPTION:
Patients are stratified into 4 early risk groups for therapy during the consolidation phase (T/early SR, T/early non-SR, pB/early non-HR, pB/early HR) and 5 risk groups for post-consolidation therapy (T/non-HR, T/HR, pB/SR, pB/MR, pB/HR). Risk stratification is based on immunophenotypic lineage, genetics of leukemic cells and treatment response on the basis of cytomorphology and methods for detection minimal residual disease.

The trial includes four randomized study questions testing experimental treatments on top of the risk-stratified standard chemotherapy backbone:

Primary study questions:

Randomization R-eHR: Early High-risk (early HR) pB-ALL defined by genetics and/or inadequate treatment response over the course of induction: Can the probability of event-free survival (pEFS) from time of randomization be improved by additional therapy with the proteasome inhibitor bortezomib during an extended consolidation treatment phase compared with standard extended consolidation?

Randomization R-HR: High-risk (HR) pB-ALL defined by genetics and/or inadequate treatment response by the end of consolidation: Can the pEFS from time of randomization be improved by a treatment concept including two cycles of post-consolidation immunotherapy with blinatumomab (15 µg/m²/d for 28 days per cycle) plus 4 doses intrathecal Methotrexate replacing two conventional highly intensive chemotherapy courses?

Randomization R-MR: Intermediate risk (MR) pB-ALL defined by genetics and intermediate MRD response: Can the probability of disease-free survival (pDFS) from time of randomization be improved by additional therapy with one cycle of post-reintensification immunotherapy with blinatumomab (15 µg/m²/d for 28 days)?

Randomization R-T: Early non-standard risk (early non-SR) T-ALL patients defined by treatment response over the course of induction: Can the pEFS from time of randomization be improved by the extension of the standard of care consolidation phase by 14 days with an increase of the consolidation cumulative doses of Cyclophosphamide, Cytarabine and 6-Mercaptopurine by 50%?

Secondary study questions:

All randomizations: Can the overall survival be improved by the treatment in the experimental arm?

All randomizations: What is the incidence of treatment-related toxicities and mortality in the experimental arm compared to the standard arm?

Randomization R-eHR: Can the MRD load after consolidation treatment be reduced by the additional treatment with bortezomib?

Randomization R-HR: Can treatment-related life-threatening complications and mortality during the intensified consolidation phase of high-risk treatment be reduced when replacing two intensive chemotherapy courses by two cycles of immunotherapy with blinatumomab?

Randomization R-HR: What is the proportion of patients with insufficient MRD response to blinatumomab as defined in the protocol as compared to the MRD response after the HR-2' block in the control arm?

Randomization R-HR: Can the MRD load after the first treatment cycle (HR 2'/blinatumomab) and the second cycle (HR-3'/blinatumomab) be reduced in the experimental arm when compared with conventional intensive chemotherapy? Randomization R-MR: What is the proportion of patients with positive MRD after reintensification Protocol II who become MRD-negative over the blinatumomab cycle compared to 4 weeks of standard maintenance therapy?

Randomization R-T: Can the MRD load after consolidation treatment be reduced by extension of the consolidation phase?

Standard-risk patients: Is the clinical outcome comparable to that obtained for standard-risk patients in study AIEOP-BFM ALL 2009?

A small subgroup of patients at very high relapse risk is eligible for allogeneic hematopoietic stem cell transplantation after the intensified consolidation therapy phase.

Patients with T-ALL and hyperleukocytosis (>=100,000/µL) and patients with CNS involvement at diagnosis (CNS3 status) are eligible for cranial irradiation with 12 Gy if age at time of irradiation is at least 4 years.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed acute lymphoblastic leukemia or
* newly diagnosed mixed phenotype acute leukemia (MPAL) meeting one of the following criteria:
* biphenotypic with a dominant T or B lineage assignment
* bilineal either with a dominant lymphoblastic population or if another reasonable rationale exists to treat the patient with an ALL-based therapy regimen
* newly diagnosed acute undifferentiated leukemia
* age < 18 years (up to 17 years and 365 days) at the day of diagnosis
* patient enrolled in a participating center
* written informed consent to trial participation and transfer and processing of data A subsequent removal from the study is only allowed if the inclusion criteria turn out not to be fulfilled or in the case of pregnancy of the patient.

Exclusion Criteria:

* Ph+ (BCR-ABL1 or t(9;22)-positive) ALL
* bilineal leukemia with a lymphoblastic and a separate non-lymphoblastic (≥ 10% of total cells) blast subset
* pre-treatment with cytostatic drugs
* glucocorticoid pre-treatment with ≥ 1 mg/kg/d for more than two weeks during the last month before diagnosis
* treatment started according to another protocol
* underlying disease that does not allow treatment according to the protocol (e.g. severe congenital heart disease, Charcot-Marie Syndrome, Ataxia-teleangiectasia…)
* ALL diagnosed as second malignancy and preceding chemotherapy and/or radiotherapy
* evidence of pregnancy or lactation period
* Sexually active adolescents not willing to use highly effective contraceptive method (pearl index <1) until 12 months after end of anti-leukemic therapy
* participation in another clinical trial except for add-on trials within the scope of supportive care approved by the sponsor
* live vaccine immunization within 2 weeks before start of protocol treatment

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5000 (Estimated)
Dates: Start 2018-07-15 (Actual); Primary Completion 2028-07-14 (Estimated); Study Completion 2028-07-14 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | Assessed up to 120 months from start of study
  Randomization R-eHR, R-HR and R-T: Time from randomization until the first event defined as follow: cytomorphological or molecular non-response (resistance to protocol treatment, considered as event at day zero), relapse, second malignancy or death from any cause. This will be called EFS time.
Disease-free survival | Assessed up to 120 months from start of study
  Randomization R-MR: Time from randomization until the first event defined as follow: Relapse, second malignancy or death from any cause. This will be called DFS time.

SECONDARY OUTCOMES:
Survival | Assessed up to 120 months from start of study
  All patients/randomizations: Time until death from any cause, starting at the same time point as the EFS/DFS.
Treatment-related mortality | Assessed up to 120 months from start of study
  Frequency and incidence of treatment-related mortality in induction or continuous complete remission
Adverse Events of interest/Serious Adverse Events | Assessed up to 120 months from start of study
  Frequency and incidence of adverse events of interest and serious adverse events in specific protocol phases, randomized arms and overall during follow-up
MRD response | Measurements of MRD response at end of randomized treatments (intended time frame 13 weeks in R-eHR/R-T, 26 weeks in R-HR, 34 weeks in R-MR).
  MRD load after the randomized treatment phases (R-eHR, R-HR, R-MR and R-T) as well as after the first/second cycle of Blinatumomab or after the HR 2'/HR 3' block (R-HR)
Proportion of patients with Blina Poor-Response | Measurements of MRD response intended after 30 weeks from individual start of treatment, assessment of proportion at 120 months from start of study
  Proportion of patients with poor MRD response to the first Blinatumomab cycle ("Blinatumomab Poor-Response") (R-HR)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schrappe, MD, Principal Investigator — Department of Pediatrics, University Hospital of Schleswig-Holstein, Campus Kiel
Locations (115):
- Australia (2):
  - Sydney Children's Hospital, Sydney
  - The Children's Hospital at Westmead, Westmead
- Austria (5):
  - Univ.Klinik für Kinder- und Jugendheilkunde Graz, Graz
  - Univ.Klinik für Kinder- und Jugendheilkunde Innsbruck, Innsbruck
  - Kepler Universitätsklinikum, Linz
  - LKH Salzburg, Salzburg
  - St. Anna Kinderspital, Vienna
- Czechia (8):
  - University Hospital Brno, Brno
  - Regional Hospital České Budějovice, České Budějovice
  - University Hospital Hradec Králové, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - University Hospital Ostrava-Poruba, Ostrava-Poruba
  - University Hospital Plzeň, Pilsen
  - University Hospital Motol, Prague
  - Masaryk´s Hospital Ústí nad Labem, Ústí nad Labem
- Germany (51):
  - Kinderklinik der med. Fakultät der RWTH, Bereich Hämatologie/Onkologie, Aachen
  - I. Klinik für Kinder u. Jugendliche, Klinikum Augsburg, Hämatologie/ Onkologie, Augsburg
  - Klinikum Berlin-Buch II. Kinderklinik, Bereich Onkologie/Allg. Pädiatrie, Berlin
  - Kinderklinik der Charité, Campus Virchow Klinikum (CVK), Abt.: Kinderhämatologie, Berlin
  - Städtisches Krankenhaus, Kinderklinik, Braunschweig
  - Klinikum Chemnitz gGmbH, Klinik für Kinder- und Jugendmedizin, Hämatologie / Onkologie, Chemnitz
  - Kliniken der Stadt Köln GmbH, Kinderkrankenhaus Riehl, Cologne
  - Med. Einrichtungen der Universität zu Köln, Klinik für Allg. Kinderheilkunde, Onkologisch-hämatologische Station, Cologne
  - Carl-Thiem-Klinikum, Kinderklinik, Abt. Hämatologie/Onkologie, Cottbus
  - Vestische Kinder- u. Jugendklinik, Universitätsklinik Witten/Herdecke, Datteln
  - Klinikum Dortmund, Klinik f. Kinder- und Jugendmedizin, Dortmund
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinik, Düsseldorf
  - Helios Klinikum Erfurt GmbH, Klinik für Kinderheilkunde, Erfurt
  - Universitaets - Kinderklinik, Erlangen
  - Universitaetsklinikum Essen, Essen
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Universitaetskinderklinik - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Klinikum der Justus-Liebig-Universität, Zentrum für Kinderheilkunde, Abt. Hämatologie/Onkologie, Giessen
  - Universitäts-Kinderklinik Päd. I, Hämatologie/Onkologie, Göttingen
  - Klinik und Poliklinik für Kinder und Jugendmedizin, Allgemeine Pädiatrie mit Poliklinik/Pädiatrische Onkologie und Hämatologie, Greifswald
  - Medizinische Hochschule Hannover, Zentrum Kinderheilkunde u. Jugendmedizin, Hanover
  - Universitäts-Kinderklinik, Päd. Onkologie, Hämatologie, und Immunologie, Heidelberg
  - Klinikum Heilbronn GmbH, Klinik für Kinderheilkunde und Jugendmedizin/Perinatalzentrum, Heilbronn
  - Gemeinschaftskrankenhaus Herdecke, Kinderabteilung, Herdecke
  - Universitaetsklinikum des Saarlandes, Homburg
  - Klinikum, der Friedrich-Schiller-Universität, Klinik für Kinder- und Jugendmedizin, Jena
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - Klinikum Kassel, Kassel
  - Klinik für Allgemeine Paediatrie, Univ.-Klinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Department für Frauen- und Kindermedizin, Abteilung für Pädiatrische Onkologie, Hämatologie und Hämostaseologie, Leipzig
  - Universität zu Lübeck, Klinik für Kinder- u. Jugendmedizin, Abt. Hämatologie/ Onkologie/Immunologie, Lübeck
  - Universitätsklinikum Magdeburg, Klinik für Päd. Hämatologie/Onkologie, Magdeburg
  - Klinikum Mannheim gGmbH, Kinderklinik, Abt. Hämatologie/Onkologie, Mannheim
  - Universitätsklinikum, Mannheim
  - Johannes Wesling Klinikum Minden, Minden
  - Städt. Krankenhaus München GmbH, Krankenhaus München-Schwabingen, Kinderklinik d. TU, München
  - Ludwig-Maximilian-Universität, Dr. von Haunersches Kinderspital, München
  - Universitäts-Kinderklinik, Päd. Hämatologie und Onkologie, Münster
  - Cnopf'sche Kinderklinik, Onkologie, Nuremberg
  - Klinikum Oldenburg gGmbH, Zentrum für Kinder- u. Jugendmedizin, (Elisabeth Kinderkrankenhaus), Oldenburg
  - Universitätsklinikum, Regensburg
  - Universitäts-Kinderklinik, Rostock
  - Asklepios-Klinik, Sankt Augustin GmbH, Sankt Augustin
  - HELIOS Kliniken Schwerin, Klinik f. Kinder-u. Jugendmedizin, Schwerin
  - Olga-Hospital, Kinderklinik, Pädiatrisches Zentrum, Abt. Hämatologie/Onkologie, Stuttgart
  - Krankenanstalt Trier, Mutterhaus der Borromaeerinnen, Pädiatrische Abteilung, Trier
  - Universitaetsklinikum Tuebingen, Tübingen
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - Stadtkrankenhaus, Kinderklinik, Wolfsburg
  - Universitaets - Kinderklinik Wuerzburg, Würzburg
- Israel (6):
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical center, Jerusalem
  - Schneider Children Medical Center of Israel, Petah Tikva
  - Sheba Medical Center Tel-Hashomer, Ramat Gan
  - Dana children hospital, Tel Aviv
- Italy (31):
  - Azienda ospedali riuniti, Ancona
  - AOUC Policlinico Bari, Bari
  - A.O. Papa Giovanni XXIII, Bergamo
  - Università di Bologna, Bologna
  - ASST Spedali Civili di Brescia, Brescia
  - Ospedale Businco, Cagliari
  - Azienda ospedaliero universitaria, Catania
  - AO Pugliese Ciaccio, Catanzaro
  - S.O. Annunziata - A. O. Cosenza, Cosenza
  - Ospedale Meyer, Florence
  - Istituto Giannina Gaslini, Genova
  - Policlinico di Modena Azienda Ospedaliero-Universitaria, Modena
  - Clinica pediatrica Fondazione MBBM, Monza
  - A.O.U. Vanvitelli, Napoli
  - AORN Santobono Pausilipon, Napoli
  - Azienda ospedaliera di Padova, Padua
  - Ospedale Civico ARNAS Civico e Di Cristina, Palermo
  - Azienda ospedaliero-universitaria di Parma, Parma
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Ospedale S. Maria della misericordia, Perugia
  - Ospedale Civile di Pescara, Pescara
  - Ospedale Santa Chiara Pisa, Pisa
  - Grande ospedale metropolitano B-M-M, Reggio Calabria
  - Ospedale infermi, Rimini
  - Fondazione Policlinico Gemelli, Roma
  - Ospedale Bambino Gesù, Roma
  - Policlinico Umberto I Università Sapienza di Roma, Roma
  - Ospedale "Casa sollievo della sofferenza", San Giovanni Rotondo
  - A.O.U. Città della salute e della scienza di Torino, Torino
  - IRCCS Burlo Garofolo, Trieste
  - AOU Verona, Verona
- Slovakia (3):
  - Klinika pediatrickej hematológie a onkológie SZU a DFNsP, Banská Bystrica
  - Comenius University Children's Hospital, Bratislava
  - Detská fakultná nemocnica Košice, Košice
- Switzerland (9):
  - Kantonsspital Aarau, Aarau
  - Universitäts-Kinderspital beider Basel, Basel
  - Ospedale San Giovanni Bellinzona, Bellinzona
  - Inselspital Bern, Bern
  - HUG Hôpitaux Universitaires de Gèneve, Geneva
  - CHUV Centre Hospitalier Universitaire Vaudois, Lausanne
  - Luzerner Kantonsspital-Kinderspital Luzern, Lucerne
  - Ostschweizer Kinderspital, Sankt Gallen
  - Universitäts-Kinderspital Zürich, Zurich

REFERENCES:
- [Derived] Tufekci O, Evim MS, Gunes AM, Celkan T, Karapinar DY, Kaya Z, Baysal B, Baytan B, Kocak U, Yilmaz S, Cinar S, Oren H. Assessment of Minimal Residual Disease in Childhood Acute Lymphoblastic Leukemia: A Multicenter Study From Turkey. J Pediatr Hematol Oncol. 2022 Mar 1;44(2):e396-e402. doi: 10.1097/MPH.0000000000002419. PMID 35129146